CLINICAL TRIAL: NCT03329664
Title: Safety and Efficacy of ex Vivo Activated and Expanded Autologous Cytokine-induced Killer Cells for Colon Cancer Patients
Brief Title: Autologous Killer Cell Therapy in Colon Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sabz Biomedicals (Industry)
Collaborators: Ministry of Health and Medical Education (Unknown); Digestive Diseases Research Institute, Tehran University of Medical Sciences, Iran (Unknown)
Responsible Party: Principal Investigator, Naser Ahmadbeigi, Doctor, Tehran University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Autologous Killer cell therapy
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Colon Cancer Stage IV
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIK Intervention plus routine treatment (Experimental): Patients who receive their routine treatment (chemotherapy, radiation therapy) + Cytokine-induced killer cell infusion
  Interventions: Biological: Cytokine-induced killer cell; Other: Chemotherapy AND/OR Radiation Therapy
- Control (Active Comparator): Patients who receive routine treatments only (chemotherapy, radiation therapy)
  Interventions: Other: Chemotherapy AND/OR Radiation Therapy

INTERVENTIONS:
Biological: Cytokine-induced killer cell — Immune-cell therapy with CIK cells
  Other Names: CIK
  Arms: CIK Intervention plus routine treatment
Other: Chemotherapy AND/OR Radiation Therapy — Routine treatments for colon cancer patients according to their stage

SUMMARY:
This study aims to evaluate the safety and efficacy of activated and expanded autologous cytokine-killer cells in controlling disease recurrence in colon cancer patients with liver metastasis. 20 patients with confirmed stage IV colon carcinoma with metastasis will be assigned into two groups. Patients in both groups will receive the same therapeutic regimen as usual. Patients in one group additionally will be treated with a single infusion of autologous killer cells that had been previously prepared from peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed colorectal cancer at stage IV
* ECOG performance status 0-2
* Adequate cardiac/renal/hepatic function
* Adequate bone marrow function (blood cell count)

Exclusion Criteria:

* Patients that have received prior chemotherapy or immune cell therapy
* Patients that have previously participated in another clinical trial
* History of positive test result for HIV, HBV, HCV, HTLV-1, syphilis
* Presence of Active infections
* Patients with immunodeficiencies, autoimmunities, or severe allergies
* Receiving immunosuppressive regimens

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-09 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Safety of administering CIK cells plus chemotherapy | one month post infusion
  Patients will be continually assessed for unexpected adverse events or unexpected early mortality 30 days post infusion
Progression-free Survival (PFS) | 2 years
  The time from treatment initiation day to first documented progressive disease or death due to disease.
Time to progression (TTP) | 2 years
  the time from randomization until cancer progression, not including death.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  The length of time that the patients are still alive at a defined period of time after treatment
Patient quality of life | each 3 months for 2 years
  Quality of patients enrolling in the study assessed using EORTC-CR29 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Naser Ahmadbeigi, Ph.D, Principal Investigator — Cell-based Therapies Research Center, Digestive Disease Research Institute, Tehran University of Medical Sciences, Tehran, Iran
Locations (1):
- Gene Therapy Research Center, Digestive Disease Research Institute, Tehran University of Medical Sciences, Tehran, Iran